CLINICAL TRIAL: NCT02383095
Title: Efficiency of Art-therapy in Psychotic Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties of recruitment
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5937
Record Dates: First submitted 2015-01-26; First posted 2015-03-09 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Art-therapy; Visual organization
MeSH Terms: conditions — Schizophrenia | interventions — Art Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Art-therapy (Experimental): 16 Art-therapy sessions
  Interventions: Behavioral: Art therapy
- Metacognitive therapy (Active Comparator): 16 Metacognitive therapy sessions
  Interventions: Behavioral: metacognitive therapy

INTERVENTIONS:
Behavioral: Art therapy
  Arms: Art-therapy
Behavioral: metacognitive therapy
  Arms: Metacognitive therapy

SUMMARY:
The main purpose of the protocol is to test the efficiency of art-therapy versus metacognitive rehabilitation on the visual perception disorders observed in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia according to DSM IV

Exclusion Criteria:

* addiction problem
* invalidating visual sensory problems
* neurological history

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in Response times between baseline and after 16 therapy sessions | Baseline and after 16 therapy sessions (up to 6 months)

SECONDARY OUTCOMES:
Change in Clinical scales (SAPS and SANS) between baseline and after 16 therapy sessions | Baseline and after 16 therapy sessions (up to 6 months)
Change in esthetic perception between baseline and after 16 therapy sessions | Baseline and after 16 therapy sessions (up to 6 months)
  Esthetic Perception Test
Change in errors in visual organization tasks between baseline and after 16 therapy sessions | aseline and after 16 therapy sessions (up to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Anne GIERSCH, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de psychiatrie, Hôpitaux Universitaires de Strasbourg, Strasbourg, France